CLINICAL TRIAL: NCT05577806
Title: Comparison of Reproductive Outcomes After Progestin-primed Ovarian Stimulation With Dydrogesterone Versus Cetrorelix to Inhibit Spontaneous Ovulation in Oocyte Donation
Brief Title: DYG Versus Cetrorelix in Oocyte Donation
Status: Completed | Type: Observational
Sponsor: Clinica de la Mujer Medicina Reproductiva, Chile (Other)
Responsible Party: Principal Investigator, Jose Antonio Moreno, MD, PhD, Clinica de la Mujer Medicina Reproductiva, Chile
Other Study IDs: PPOS-DU-OD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Infertility, Female; Fertility Disorders
Keywords: Gonadotrophin-releasing hormone (GnRH) analogues; Ovarian stimulation; Oocyte donation; Progestin-primed ovarian stimulation; Dydrogesterone
MeSH Terms: conditions — Infertility, Female | interventions — Dydrogesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DYG: oocyte donors undergoing controlled ovarian stimulation in a progestin-primed ovarian stimulation protocol with DYG protocol (20mg/day)
  Interventions: Drug: Dydrogesterone
- Cetrorelix: oocyte donors undergoing controlled ovarian stimulation in a GnRH antagonist protocol with cetrorelix (0.25 mg/day) from Day 7 or since a leading follicle reached 14 mm

INTERVENTIONS:
Drug: Dydrogesterone — progestin primed ovarian stimulation
  Groups: DYG

SUMMARY:
Prospective controlled study to assess the reproductive outcomes of OD recipients in which the donors were subjected to the DYG protocol (20mg/day) compared with those subjected to the short protocol with cetrorelix (0.25 mg/day) from Day 7 or since a leading follicle reached 14 mm. The OD cycles were triggered with triptoreline acetate and the trigger criterion was ≥3 follicles of diameter >18mm.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors between 21 and 30 years old, with regular menstrual cycles (24-35 d) and a body mass index (BMI) between 18 and 28 kg/m2 without any relevant personal or family history

Exclusion Criteria:

* AMH less than 3 ng/dL
* A positive screening for sexually transmitted diseases

Ages: 21 Years to 30 Years | Sex: Female
Age Groups: Adult
Study Population: Oocyte donors undergoing controlled ovarian stimulation
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate per transfer | 40 weeks after ET
Clinical pregnancy per transfer | 12 weeks after ET
Miscarriage rate | 12 weeks after ET

SECONDARY OUTCOMES:
Number of oocytes retrieved | at time of oocyte retrieval
Number of mature oocytes | 1 day after IVF
Number of fertilized oocytes | 1 day after IVF
Number of blastocists | 5-6 days after OPU

IPD SHARING:
Plan to Share IPD: Undecided